CLINICAL TRIAL: NCT01150838
Title: Propofol for Pediatric Tracheal Intubation With Deep Anesthesia During Sevoflurane Induction: Dosing According to Elapsed Time for Two Age Groups,IRB-HSR# 13666
Brief Title: Propofol for Pediatric Tracheal Intubation With Deep Anesthesia During Sevoflurane Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, George Politis, MD, Attending Anesthesiologist, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 13666
Record Dates: First submitted 2010-06-02; First posted 2010-06-28 (Estimated); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Anesthesia Intubation Complication
Keywords: intubation of children without neuromuscular blockade
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Intervention Model Description: This is a single study with 6 parallel groups as noted in the description. With Dixon's Up and Down Method for determining a 50th percentile of a dichotomous outcome, the number of patients required is not known prior to starting a study. Data from Paul and Fisher demonstrated that 6 "crossovers" (change in the dichotomous outcome from one patient to another, indicating change from increasing the dose of the study drug to decreasing it, or visa-versa). When choosing a meaningful starting point near the 50th percentile, the number required is typically 15-20 patients. With 6 study groups, the estimated number of patients required would be 90-120. Please Note: This is not a study where one can perform a power analysis and determine a required N.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Propofol administration (Experimental): For each of the 6 groups, propofol 2 mg/kg will be administered to first subject. The propofol dose will move separately for each of the 6 groups, and be increased by 0.3 mg/kg for the next subject if intubation score is "not excellent" and decreased by 0.3 mg/kg if intubation score is "excellent". This dosing scheme will be continued until there are 6 "crossovers" as described above.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — Initial dose: Propofol 2 mg/kg, then dose changes separately based on the last subject in the same age group and sevo time range

SUMMARY:
The purpose of this study is to determine the amount of propofol required to achieve 50% of patients obtaining a perfect ("excellent") intubation score of 5 on the Steyn modification of the Helbo-Hansen Intubation Score, when placing a tracheal tube in children 1-6 years and 6-12 years (division of age groups at 6th birthday) of age, under a specific induction and ventilation sequence as specified in this study design.

DETAILED DESCRIPTION:
The practice of tracheal intubation of children without neuromuscular blockade (TIWNB) is widespread in pediatric anesthesia practices. There are several different methods reported for TIWNB, most of which involve administration of an inhaled anesthetic in combination with an intravenous adjunctive medication. The technique of administering propofol IV, immediately after IV placement, after a sevoflurane induction is perhaps the most popular method for pediatric TIWNB in the United States and worldwide (personal communication, and personal practice of this technique). At the time this study was proposed, nobody had studied this technique, and therefore nobody had quantified the amount of propofol needed in this context, or considered that the amount may differ according to the time sevoflurane has been administered at the moment propofol is given. This study divides patients into two age categories, with the first age group starting at the 1 year birthday and going up to the 6th year birthday, and the second age group going from the 6th year birthday up to the 12th birthday. The study also divides participants according to time that they have received sevoflurane from the start of anesthetic induction until intravenous access is achieved and propofol immediately administered. That amount of time varies in clinical practice due to variable difficulty obtaining pediatric intravenous access, and the amount of propofol may vary according to the amount of sevoflurane administered (time administered) because depth of anesthesia will increase with increasing duration of sevoflurane administration. The purpose of this study is to determine for both age groups the amount of propofol required to achieve 50% of patients obtaining a perfect intubation score of 5 on the Steyn modification of the Helbo-Hansen Intubation Score (HH Score), when placing a tracheal tube after various time periods of administration of sevoflurane. The 3 different time windows for sevoflurane administration prior to the propofol bolus will be 2-4 minutes, 4-6 minutes, and 6-8 minutes, starting the time clock at the start of anesthetic induction and ending at the moment the propofol is given. The study therefore has 6 separate groups (2 age groups x 3 time period groups) each of which utilizes a Dixon's Up and Down Method, moving up or down on the amount of propofol administered according to the result of the previous patient in each group (HH Score of 5 labeled "excellent intubation" indicates allocation of predetermined (0.3 mg/kg) incrementally smaller amount of propofol and >5 labeled as "not-excellent intubation" an increase of 0.3 mg/kg of propofol. Linear regression will be used for each of the 6 groups to determine the amount of propofol required to achieve 50% perfect intubation, with 95% confidence intervals also calculated.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent / assent
* Ages 1-11 years (12 - 132 months)
* American Society of Anesthesiology (ASA) physical status 1 or 2, which implies that the patient has no comorbidity that limits daily function.
* Scheduled for non-emergent surgery/ procedure under general anesthesia in which the anesthesia team intends to place an endotracheal tube
* Expected routine intubation according to physical exam and history
* Weight under 50 kg

Exclusion Criteria:

* Requires neuromuscular blocking agents
* Emergent surgery / procedure
* Expected difficult intubation
* ASA physical status 3 or 4
* Weight over 50 kg
* Age under 12 months or over 132 months
* Allergy to study drugs to be used

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George D Politis, MD, Principal Investigator — UVA Department of Anesthesiology
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Politis GD, Tobin JR, Morell RC, James RL, Cantwell MF. Tracheal intubation of healthy pediatric patients without muscle relaxant: a survey of technique utilization and perceptions of safety. Anesth Analg. 1999 Apr;88(4):737-41. doi: 10.1097/00000539-199904000-00009. PMID 10195514
- [Background] Politis GD, Frankland MJ, James RL, ReVille JF, Rieker MP, Petree BC. Factors associated with successful tracheal intubation of children with sevoflurane and no muscle relaxant. Anesth Analg. 2002 Sep;95(3):615-20, table of contents. doi: 10.1097/00000539-200209000-00022. PMID 12198047
- [Background] Simon L, Boucebci KJ, Orliaguet G, Aubineau JV, Devys JM, Dubousset AM. A survey of practice of tracheal intubation without muscle relaxant in paediatric patients. Paediatr Anaesth. 2002 Jan;12(1):36-42. doi: 10.1046/j.1460-9592.2002.00727.x. PMID 11849573
- [Background] Blair JM, Hill DA, Bali IM, Fee JP. Tracheal intubating conditions after induction with sevoflurane 8% in children. A comparison with two intravenous techniques. Anaesthesia. 2000 Aug;55(8):774-8. doi: 10.1046/j.1365-2044.2000.01470.x. PMID 10947692
- [Background] Dixon WJ. Quantal response to variable experimentation: the up-and-down method. In: McArthur JW, Colton T, eds. Statistics in Endocrionolgy. Cambridge: MIT Press, 1967: 251-264.
- [Background] Viby-Mogensen J, Engbaek J, Eriksson LI, Gramstad L, Jensen E, Jensen FS, Koscielniak-Nielsen Z, Skovgaard LT, Ostergaard D. Good clinical research practice (GCRP) in pharmacodynamic studies of neuromuscular blocking agents. Acta Anaesthesiol Scand. 1996 Jan;40(1):59-74. doi: 10.1111/j.1399-6576.1996.tb04389.x. PMID 8904261
- [Background] Steyn MP, Quinn AM, Gillespie JA, Miller DC, Best CJ, Morton NS. Tracheal intubation without neuromuscular block in children. Br J Anaesth. 1994 Apr;72(4):403-6. doi: 10.1093/bja/72.4.403. PMID 8155439
- [Background] Paul M, Fisher DM. Are estimates of MAC reliable? Anesthesiology. 2001 Dec;95(6):1362-70. doi: 10.1097/00000542-200112000-00014. PMID 11748393
- [Background] Hansen D, Schaffartzik W, Dopjans D, Heitz E, Striebel HW. Halothane-propofol anaesthesia for tracheal intubation in young children. Br J Anaesth. 1997 Apr;78(4):366-9. doi: 10.1093/bja/78.4.366. PMID 9135352
- [Background] Min SK, Kwak YL, Park SY, Kim JS, Kim JY. The optimal dose of remifentanil for intubation during sevoflurane induction without neuromuscular blockade in children. Anaesthesia. 2007 May;62(5):446-50. doi: 10.1111/j.1365-2044.2007.05037.x. PMID 17448054
- [Background] Nishina K, Mikawa K, Shiga M, Maekawa N, Obara H. Oral clonidine premedication reduces minimum alveolar concentration of sevoflurane for tracheal intubation in children. Anesthesiology. 1997 Dec;87(6):1324-7. doi: 10.1097/00000542-199712000-00010. PMID 9416716
- [Background] Inomata S, Nishikawa T. Determination of end-tidal sevoflurane concentration for tracheal intubation in children with the rapid method. Can J Anaesth. 1996 Aug;43(8):806-11. doi: 10.1007/BF03013033. PMID 8840060
- [Background] Inomata S, Yamashita S, Toyooka H, Yaguchi Y, Taguchi M, Sato S. Anaesthetic induction time for tracheal intubation using sevoflurane or halothane in children. Anaesthesia. 1998 May;53(5):440-5. doi: 10.1046/j.1365-2044.1998.00338.x. PMID 9659016
- [Background] Mencke T, Echternach M, Kleinschmidt S, Lux P, Barth V, Plinkert PK, Fuchs-Buder T. Laryngeal morbidity and quality of tracheal intubation: a randomized controlled trial. Anesthesiology. 2003 May;98(5):1049-56. doi: 10.1097/00000542-200305000-00005. PMID 12717124
- [Background] Vakkuri A, Yli-Hankala A, Sarkela M, Lindgren L, Mennander S, Korttila K, Saarnivaara L, Jantti V. Sevoflurane mask induction of anaesthesia is associated with epileptiform EEG in children. Acta Anaesthesiol Scand. 2001 Aug;45(7):805-11. doi: 10.1034/j.1399-6576.2001.045007805.x. PMID 11472278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at an outpatient surgery center
Pre-assignment Details: Four patients dropped out due to protocol violations or ended up outside the three time periods by the time IV access obtained.
Groups:
- Age 1-6 Years, Time 2-4 Minutes of Sevoflurane Until Propofol Administration; Age 1-6 Years, Time 4-6 Minutes of Sevoflurane Until Propofol Administration; Age 1-6 Years, Time 6-8 Minutes of Sevoflurane Until Propofol Administration; Age 6-11 Years, Time 2-4 Minutes of Sevoflurane Until Propofol Administration; Age 6-11 Years, Time 4-6 Minutes of Sevoflurane Until Propofol Administration; Age 6-11 Years, Time 6-8 Minutes of Sevoflurane Until Propofol Administration: Propofol 2 mg/kg administered to first subject. Dose will be increased by 0.3 mg/kg for the next subject if intubation score is "not excellent". Dose will be decreased by 0.3 mg/kg if intubation score is "excellent". This dosing scheme will be continued until at least 6 "crossovers" are achieved.
Period: Overall Study
Arm/Group | Age 1-6 Years, Time 2-4 Minutes of Sevoflurane Until Propofol Administration | Age 1-6 Years, Time 4-6 Minutes of Sevoflurane Until Propofol Administration | Age 1-6 Years, Time 6-8 Minutes of Sevoflurane Until Propofol Administration | Age 6-11 Years, Time 2-4 Minutes of Sevoflurane Until Propofol Administration | Age 6-11 Years, Time 4-6 Minutes of Sevoflurane Until Propofol Administration | Age 6-11 Years, Time 6-8 Minutes of Sevoflurane Until Propofol Administration
Started | 19 | 26 | 24 | 15 | 16 | 2
Completed | 19 | 26 | 24 | 15 | 16 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Two patients in Age 6-11 years, 6-8 minutes, did not appear in baseline analysis population due to inadequate numbers collected in that age group and time range to be able to analyze; IV access always achieved earlier that 6 minutes due to ease of IV access.
Groups:
- Age 1-6 Years, Time 2-4 Minutes of Sevoflurane Until Propofol Administration; Age 1-6 Years, Time 4-6 Minutes of Sevoflurane Until Propofol Administration; Age 1-6 Years, Time 6-8 Minutes of Sevoflurane Until Propofol Administration; Age 6-11 Years, Time 2-4 Minutes of Sevoflurane Until Propofol Administration; Age 6-11 Years, Time 4-6 Minutes of Sevoflurane Until Propofol Administration: Propofol 2 mg/kg administered to first subject. Dose will be increased by 0.3 mg/kg for the next subject if intubation score is "not excellent". Dose will be decreased by 0.3 mg/kg if intubation score is "excellent". This dosing scheme will be continued.
  propofol: Initial dose: Propofol 2 mg/kg, then dose changes separately based on the last subject in the same age group and sevo time range
- Total: Total of all reporting groups
Arm/Group | Age 1-6 Years, Time 2-4 Minutes of Sevoflurane Until Propofol Administration | Age 1-6 Years, Time 4-6 Minutes of Sevoflurane Until Propofol Administration | Age 1-6 Years, Time 6-8 Minutes of Sevoflurane Until Propofol Administration | Age 6-11 Years, Time 2-4 Minutes of Sevoflurane Until Propofol Administration | Age 6-11 Years, Time 4-6 Minutes of Sevoflurane Until Propofol Administration | Total
Number analyzed (Participants) | 19 | 26 | 24 | 15 | 16 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 26 | 24 | 15 | 16 | 100
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — No sex/gender data was collected. Population: No sex/gender data was collected.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 26 | 24 | 15 | 16 | 100

OUTCOME MEASURES:

1. Primary Outcome: Estimated Propofol Doses Producing 50% Excellent Intubation Conditions
Description: Logistic regression utilized to measure the amount of propofol to obtain 50% excellent intubation conditions for each age/time group.
  The quality of tracheal intubation will be graded according to the Steyn modification of the Helbo-Hansen scoring system for tracheal intubation, which includes evaluation of ease of laryngoscopy, position of the vocal cords, coughing, jaw relaxation and movement of limbs, each evaluated on a 1-4 scale, with 1 being the best possible condition and 4 the worst. The intubation conditions will be classified as either excellent or not-excellent. "Excellent" will be defined as a total score of 5, a score of 1 for each category, and "not-excellent" will be a total score of 6-20, meaning a score of >1 in any category. While the outcome measure of each intubation is "excellent" or "not excellent", the overall outcome being generated is the amount of propofol in mg/kg required for 50% excellent intubation score.
Time Frame: Amount of time it takes to intubate each patient; approximate time is 15-45 seconds
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mg/kg
Arm/Group | Age 1-6 Years, Time 2-4 Minutes of Sevoflurane Until Propofol Administration | Age 1-6 Years, Time 4-6 Minutes of Sevoflurane Until Propofol Administration | Age 1-6 Years, Time 6-8 Minutes of Sevoflurane Until Propofol Administration | Age 6-11 Years, Time 2-4 Minutes of Sevoflurane Until Propofol Administration | Age 6-11 Years, Time 4-6 Minutes of Sevoflurane Until Propofol Administration
Number analyzed (Participants) | 19 | 26 | 24 | 15 | 16
mg/kg | 1.48 [0.8 to 2.03] | 0.00 [0.00 to 0.38] | 0.07 [0.00 to 0.68] | 2.35 [1.97 to 2.45] | 2.33 [1.59 to 2.45]

ADVERSE EVENTS:
Time Frame: Adverse events data was collected only on day 0, starting at the time of anesthetic induction through the remaining time in the operating room, and through the recovery period, until time of discharge from the post-anesthetic care unit.
Description: Patients in this study are intubated with a method used by all the participating anesthesiologists, regardless of the patient's participation in this study. The difference with study participation is that the amount of propofol chosen for study participants is determined by protocol rather than by the anesthesiologist, and this PI believes the protocol is more likely to drive the dose to achieve adequate depth for intubation, thereby reducing All-Cause Mortality by decreasing laryngospasm.
Groups:
- Propofol Administration: Propofol 2 mg/kg administered to first subject. Dose will be increased by 0.3 mg/kg for the next subject if intubation score is "not excellent". Dose will be decreased by 0.3 mg/kg if intubation score is "excellent". This dosing scheme will be continued.
Arm/Group | Propofol Administration
All-Cause Mortality (participants affected / at risk) | 0/106
Serious Adverse Events (participants affected / at risk) | 0/106
Other Adverse Events (participants affected / at risk) | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes